CLINICAL TRIAL: NCT01149616
Title: Effects of Perioperative Intravenous Dexamethasone on Pain in Out Patient Knee Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: investigators changed jobs, no longer affiliated with institution
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lauren J. Fisher, Attending Physician, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P000345
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Post Operative Pain; Nausea
MeSH Terms: conditions — Pain, Postoperative; Nausea | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Dexamethasone 8mg iv x 1
  Interventions: Drug: Dexamethasone 8mg iv x1
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexamethasone 8mg iv x1 — Dexamethasone 8mg iv x1
  Arms: Intervention
Drug: placebo — 2 ml normal saline IV x1
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the opiate sparing effects of intravenously administered dexamethasone in outpatient knee surgery. Dexamethasone is a glucocorticoid with well known antiemetic effects. However, the analgesic effects of dexamethasone have not been adequately researched. Following surgery, patients are typically discharged home with PO opiates to manage post-operative pain. The investigators believe that by using VAS (Visual Analog Scale) for Pain the investigators can show that a single dose of dexamethasone can reduce pain scales and opiate consumption post-operatively, on Post Operative Day (POD 1) when compared to placebo.

DETAILED DESCRIPTION:
Findings of Modest improvement in pain scores and postoperative nausea at 24 hours with Dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing ambulatory knee arthroscopy surgery
* Must provide phone contact number and agree to phone followup on post operative day 1

Exclusion Criteria:

* Patients with major systemic disease
* Allergy or intolerance to study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Fisher, DO, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2010
Groups:
- Placebo: placebo
  placebo: placebo administered IV x1
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 26 | 25 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Post Operative VAS Pain Scale
Description: Patients were instructed to select a number between zero and ten to indicate the degree of pain they experience (zero being no pain and ten being the worst pain they could imagine). Therefore, ten is worse than zero.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 1.88 (0.3) | 3.73 (0.5)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.007, ANOVA

2. Secondary Outcome: Amount of Postop Narcotic Usage
Description: Patients were requested to record the number of prescribed oral analgesic (oxycodone 5 mg/aceteminophen 325 mg) tablets taken for the first 24 hours following discharge
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: number of tablets
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 41 | 41
number of tablets | 1 [1 to 2] | 2 [2 to 4]
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.006, ANOVA

3. Secondary Outcome: Postop Nausea
Description: NRS scale 0-10 for nausea. Zero indicates no nausea, Ten indicates the worst nausea imagined.
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 0 [0 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.05, ANOVA — P value was calculated, and threshold for significance calculated at less than or equal to 0.05

ADVERSE EVENTS:
Groups:
- Placebo: placebo
  placebo: placebo administered 2 ml normal saline IV x1
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No